CLINICAL TRIAL: NCT05715489
Title: Evaluation of the Results of Laparoscopic Pectopexy Surgery Without Using Mesh
Brief Title: Pectopexy Surgery Without Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Süleyman Salman, Associate Professor, Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpaşaTREHy
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with pelvic organ prolapse undergone pectopexy without using mesh (Other)
  Interventions: Procedure: Comparison of pre and postoperative POP-Q values of the patients; Procedure: Comparison of pre and postoperative PISQ-12 scores of the patients

INTERVENTIONS:
Procedure: Comparison of pre and postoperative POP-Q values of the patients — Pectopexy Without Using Mesh will be applied to the patients and POP-Q values will be compared pre and postoperatively
Procedure: Comparison of pre and postoperative PISQ-12 scores of the patients — Pectopexy Without Using Mesh will be applied to the patients and PISQ-12 scores will be compared pre and postoperatively

SUMMARY:
it is aimed to examine the effect of laparoscopic pectopexy surgery without mesh on Pelvic Organ Prolapse Measurement (POP-Q) and quality of life of the patient.

DETAILED DESCRIPTION:
Every gynecological patient with prolapse is evaluated with POP-Q staging. The POP-Q staging to be performed before the laparoscopic pectopexy operation without mesh (performed by using non-melting sutures with natural tissue repair) performed on the patients will be compared with the POP-Q staging that will be performed 6 months after the operation. In addition, the quality of life of patients before and 6 months after the operation will be compared with the incontinence quality of life scale questionnaire of Pelvic Organ Prolapse / Incontinence Sexual Questionnaire (PISQ-12).

ELIGIBILITY:
Inclusion Criteria:

* having pelvic organ prolapse greater than stage 2 according to POP-Q evaluation system
* being sexually active

Exclusion Criteria:

* Disease requiring chronic steroid use
* Asthma
* Having chronic obstructive pulmonary disease
* Having malignancy,
* Having metabolic and rheumatological diseases that impair tissue healing, such as scleroderma

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Pre and post operative assessment of POP-Q measurements | 2 year
  POP-Q values of patients before and after laparoscopic pectopexy surgery without mesh on Pelvic Organ Prolapse will be compared.
Pre and post operative assessment of Pelvic Organ Prolapse / Incontinence Sexual | 2 year
  Units on a scale of the patients obtained with Pelvic Organ Prolapse / Incontinence Sexual Questionnaire (PISQ-12) will be compared before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Salman, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes